CLINICAL TRIAL: NCT03006042
Title: Pharmacokinetics of Bupivacaine Following Bilateral Ultrasound-guided Transversus Abdominis Plane Block for Cesarean Section
Brief Title: Pharmacokinetics of BPV Following Bilateral US-guided TAP Block for C-section
Status: Completed | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, MD, assistant professor, University Tunis El Manar
Other Study IDs: UTEM BPV
Record Dates: First submitted 2016-12-20; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Anesthesia; Adverse Effect; Cesarean Section; Transversus Abdominis Plane Block
Keywords: bupivacaine; local anaesthetics; cesarean section; transversus abdominis plane block; toxicity; ultrasound guidance; QTc interval
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bupivacaine

SUMMARY:
The transversus abdominis plane block (TAP block) is an effective method of postoperative pain management after cesarean section (C-section). Up to now, there are no data available about bupivacaine (BPV) plasma levels after TAP block in adults. In the current study, the investigators aimed to assess BPV pharmacokinetic parameters after ultrasound-guided TAP block using BPV in parturients undergoing C-section and to report its effects on corrected QT interval.

DETAILED DESCRIPTION:
The investigators led a prospective observational study in pregnant women undergoing elective C-section under spinal anesthesia (SA) using 10 mg of hyperbaric BPV. After surgery, they received bilateral ultrasound-guided TAP block with 50 mg of BPV in each side. Venous blood samples were collected immediately before and at 10, 30, 45, 60, 90, 120, 180, 240, 720 and 1440 minutes after both TAP blocks. The investigators used high performance liquid chromatography (HPLC) to measure BPV total plasma concentrations. Mean BPV area under the curve (AUC) was calculated from 0 to 24 hours according to the linear trapezoidal rule. Mean peak of total BPV plasma concentration (Cmax) and time to reach the peak (Tmax) were recorded. Electrocardiographic (ECG) recordings were also repeated at 1, 2, 3 and 4 hours to investigate the effect of BPV on corrected QT (QTc) intervals. Data were computed using SPSS 20®. Quantitative data were expressed as means ± SD. Qualitative data were expressed as percentages.

ELIGIBILITY:
Inclusion Criteria:

ASA physical status I-II pregnant women scheduled for elective C-section with Pfannenstiel incision under Spinal anesthesia

Exclusion Criteria:

* ASA physical status > II,
* known allergy to local anesthetics,
* body mass index (BMI) more than 40 kg/m²,
* coagulation disorders,
* neurologic or neuromuscular disease,
* significant liver or renal dysfunction,
* electrolyte disturbances,
* heart arrhythmias,
* corrected QT (QTc) interval> 0.47s
* patients taking drugs that may prolong QT interval.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: After obtaining approval by the institute ethics committee and having written informed consent signed on the day of surgery, 17 American Society of Anesthesiologists (ASA) physical status I-II pregnant women aged between 20 and 40 years scheduled for elective C-section with Pfannenstiel incision, under SA, were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Total venous plasma concentration of BPV | Immediately before and at 10, 30, 45, 60, 90, 120, 180, 240, 720 and 1440 minutes after both TAP blocks.

SECONDARY OUTCOMES:
corrected QT interval | at 1, 2, 3 and 4 hours after TAP blocks

IPD SHARING:
Plan to Share IPD: No